CLINICAL TRIAL: NCT06712134
Title: The Factors Associated 30-day Mortality After Perioperative Cardiac Arrest in Adults Undergoing Non-cardiac Surgery: A 7-year Observational Study From a Tertiary Care University Hospital
Brief Title: The Factors Associated 30-day Mortality After Perioperative Cardiac Arrest in Adults Undergoing Non-cardiac Surgery.
Status: Completed | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Pattrapun Wongsripuemtet, Instructor Anesthesiologist, Siriraj Hospital
Other Study IDs: 321/2022
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Arrest; Perioperative Complication
Keywords: Critical care; Perioperative cardiac arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Perioperative cardiac arrest (PCA) in patients undergoing noncardiac surgery is a rare but potentially catastrophic event associated with high mortality. Several studies have highlighted the factors contributing to PCA in the surgical population. However, information on outcomes after PCA among the surgical population is still limited. Our study aims to identify the incidence of PCA, 30-days mortality and the factors associated with PCA and 30-day mortality after PCA in adults undergoing non-cardiac surgery

ELIGIBILITY:
Inclusion Criteria:

* patients aged> 18 years old
* history of perioperative cardiac arrest
* non- cardiac surgery

Exclusion Criteria:

* did not receive cardiopulmonary resuscitation (CPR) during PCA
* incomplete data regarding 30-day mortality were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >eighteen years that had non-cardiac surgery under anesthesia and a history of PCA between January 2015 and December 2021 were eligible for inclusion. Patients with a do not resuscitate (DNR) order, who did not receive cardiopulmonary resuscitation (CPR) during PCA, or with incomplete data regarding 30-day mortality were excluded. PCA was defined as the absence of mechanical heart function (determined by a central pulse) and loss of effective circulation between the administration of anesthesia until 24 hours after surgery
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
incidence of 30 days mortality after perioperative cardiac arrest | 30 days
  incidence of 30 days mortality after perioperative cardiac arrest